CLINICAL TRIAL: NCT05701215
Title: Venetoclax After TKI to Target Persisting Stem Cells in CML
Acronym: VARIANT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Ernst, PD Dr. med. (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Thomas Ernst, PD Dr. med., Principal Investigator, University of Jena
Organization: University of Jena (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VARIANT; 2022-003069-39 (EudraCT Number)
Record Dates: First submitted 2022-10-26; First posted 2023-01-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Venetoclax (Experimental): Venetoclax will be taken orally once daily (400 mg) for 12 months after stop of TKI
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be taken orally once daily (400 mg) for 12 months

SUMMARY:
There is currently no available treatment, capable to increase the rate of sustained deep molecular remissions after TKI discontinuation in CML. Venetoclax could be such a drug. The study will provide unprecedented biological insights on the effects of venetoclax in controlling minimal residual stem cell disease induced by long-term prior TKI therapy. If the study would be positive, the findings could become practice changing for patients in deep molecular remission under TKI and willing to tolerate a temporary additional treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of chronic phase CML with cytogenetic confirmation of the Philadelphia (Ph) chromosome
2. Ph negative cases or patients with variant translocations who are BCR::ABL1 positive in multiplex PCR are also eligible
3. Typical b2a2 and/or b3a2 BCR::ABL1 transcripts
4. Subject must be ≥ 18 years of age
5. Stored DNA from initial diagnosis (prior TKI treatment) for BCR::ABL1 breakpoint analysis
6. BCR::ABL1 transcript level according to the international scale (IS) of MR4 or better which has been confirmed three times within the past 13 months and was assessed by an IS-certified reference laboratory, such as of the University Jena or another MR4-certified laboratory in Germany
7. At least 3 years of TKI therapy
8. Patients who failed to discontinue TKI in a prior discontinuation attempt are still eligible if they fulfill criteria 6 after retreatment with TKI
9. WHO performance status 0-2
10. Adequate end organ function as defined by:

    * Total bilirubin (TBL) < 3 x Upper Limit of Normal (ULN); patients with Gilbert's syndrome may only be included if TBL ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN,
    * Creatinine Clearance (CrCl) ≥ 30 millilitres per minute (mL/min) as calculated using Cockcroft-Gault formula, Serum lipase ≤ 1.5 x ULN. For serum lipase > ULN 1.5 x ULN, value must be considered not clinically significant and not associated with risk factors for acute pancreatitis.
11. Patients must have the following laboratory values within normal limits or corrected to within normal limits with supplements:

    * Potassium (potassium increase of up to 6.0 mmol/L is acceptable if associated with CrCl ≥ 90 mL/min),
    * Total calcium (corrected for serum albumin); (calcium increase of up to 12.5 mg/dl or 3.1 mmol/L is acceptable if associated with CrCl ≥ 90 mL/min),
    * Magnesium (magnesium increase of up to 3.0 mg/dL or 1.23 mmol/L if associated with CrCl ≥ 90 mL/min),
    * For patients with mild to moderate renal impairment (CrCl ≥ 30 mL/min and <90 mL/min) - potassium, total calcium (corrected for serum albumin) and magnesium should be within normal limits or corrected to within normal limits with supplements.
12. Women of childbearing age must use a highly effective method of contraception while using venetoclax. Women using hormonal contraceptives should also use a barrier method.
13. Negative pregnancy test in women of childbearing potential
14. Subject must voluntarily sign and date an informed consent

Exclusion Criteria:

1. Concomitant use of strong CYP3A-Inhibtors (e.g., itraconazole, ketoconazole, posaconazole, voriconazole, clarithromycin, ritonavir) is contraindicated
2. Concomitant use of moderate CYP3A-Inhibitors (e.g., ciprofloxacin, diltiazem, erythromycin, fluconazole, verapamil) should be avoided.
3. Grapefruit products, Seville oranges, and starfruit (carambola) should be avoided during treatment with venetoclax as they contain inhibitors of CYP3A
4. Concomitant use of venetoclax with P-gp and BCRP inhibitors
5. Concomitant use of venetoclax with strong CYP3A inducers (e.g., carbamazepine, phenytoin, rifampin) or moderate CYP3A inducers (e.g., bosentan, efavirenz, etravirine, modafinil, nafcillin) should be avoided
6. Concomitant use of preparations containing St. John´s wort
7. Patients with severe renal impairment (Crea-Clearance < 30 ml/min) or on dialysis
8. Patients with severe hepatic impairment
9. Patients who are pregnant or breast feeding, or females of reproductive potential not employing an effective method of birth control. Female patients must agree to employ an effective barrier method of birth control throughout the study and for and for at least 30 days after ending venetoclax treatment
10. Known impaired cardiac function
11. Impaired gastrointestinal function or disease that may alter the absorption of study drug
12. Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
13. Active or uncontrolled infections at the time of enrolment
14. Known HIV sero-positivity or known active hepatitis B or C infection (HIV testing is not required)
15. Participation in another clinical study with other investigational drugs within 14 days prior to enrolment
16. Any medical, mental, psychological or psychiatric condition that in the opinion of the investigator would not permit the patient to complete the study or understand the patient information
17. Subject has acute leukemia
18. Subject has known active CNS involvement.
19. Hypersensitivity to venetoclax or any component of the formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
stem cell change | at 6 months and 12 months after start of Venetoclax
  Reduction of BCR::ABL1 stem cells measured by quantitative genomic PCR in bone marrow after venetoclax administration.

SECONDARY OUTCOMES:
European Organisation for Research and Treatment of Cancer - Quality of Life C30 - Questionnaire | at 6 months and 12 months after start of Venetoclax
  compared to baseline with EORTC-QLQ C30 - Questionnaire (Score from 1 to 4; 1 better, 4 worse)
Kinetics of BCR::ABL1-transcript expression | monthly after start of Venetoclax until month 12
  Kinetics of typical BCR::ABL1 transcript level over time after Tyrosine kinase stop
Overall survival (OS) | monthly after start of Venetoclax until month 12
  defined as the time between the date of enrollment and the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ernst, Prof. Dr., Principal Investigator — University Hospital Jena
Locations (2):
- Germany (2):
  - Uniklinik der RWTH Aachen, Aachen
  - Universitätsklinikum Jena, Jena

IPD SHARING:
Plan to Share IPD: No